CLINICAL TRIAL: NCT01056523
Title: A Phase I/II Study of Ribavirin and Low-dose Cytarabine Arabinoside (Ara-C) in Acute Myeloid Leukemia (AML) M4 and M5 Subtypes, and AML With High eIF4E Expression
Brief Title: Use of Ribavirin and Low Dose Ara-C to Treat Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Sarit Assouline, Principal Investigator, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ribavirin-002
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Ribavirin; Arabinofuranosylcytosine Triphosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ribavirin-Cytarabine arabinoside (Experimental): Ribavirin will be given orally bid according to a dose escalation scheme daily for 28 days of a 28 day cycle Cytarabine arabinoside will be given 20 mg sc bid days 1 to 10 of a 28 day cycle
  Interventions: Drug: Ribavirin; Drug: Cytarabine arabinoside

INTERVENTIONS:
Drug: Ribavirin — Dose level 1 = 1000 mg po BID/ Dose level 2 = 1400 mg po BID/ Dose level 3 = 1800 mg po BID
Drug: Cytarabine arabinoside — Previous cohorts at 20 mg bid days 1 to 10 of every 28 day cycle. Dosage modified to 10 mg bid days 1 to 10 of every 28 day cycle for more recent cohorts.
  Other Names: Ara-C

SUMMARY:
The purpose of the study is to determine the maximum tolerated dose of ribavirin, when given in combination with low-dose ara-C and to determine if it is safe and well-tolerated in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
Primary Objectives

In the Phase I portion of this study, we will determine the maximum tolerated dose and recommended phase II dose (RP2D) of ribavirin and low-dose ara-C. The primary objective of the Phase II portion of the study is to determine the overall response rate, including the complete remission (CR), complete remission with incomplete blood count recovery (CRi), partial remission (PR) or blast response (BR), to therapy with ribavirin and low dose ara-C at the RP2D.

STUDY DESIGN AND DURATION

This is a multicentre, open-label, single arm Phase I/II study of oral ribavirin and low-dose ara-C for patients with AML M4/M5 or AML with high expression of eIF4E, who have relapsed or refractory disease, or who are not suitable candidates for induction chemotherapy. This study will determine the recommended phase II dose and will evaluate efficacy. Correlative studies will be included to assess relevant molecular targets.

ELIGIBILITY:
Inclusion Criteria:

* The following patients with acute myeloid leukemia (AML) are eligible:

  * De novo AML M4 or M5 FAB subtype or high eIF4E.
  * Secondary AML after a myelodysplastic syndrome (MDS) or a myeloproliferative disorder (not chronic myelogenous leukemia), if M4 or M5 FAB subtype or high eIF4E.
  * Therapy-related AML if M4 or M5 FAB subtype or high eIF4E.
  * CML blast crisis if they have failed imatinib and at least one other tyrosine kinase inhibitor.
* All patients must have failed primary therapy (defined as two induction chemotherapies), have relapsed, or are not suitable candidates for intensive induction chemotherapy.
* Patients who have a dry aspirate or extramedullary disease only are eligible for this study if they have a pre-treatment marrow or tissue biopsy demonstrating AML M4 or M5 subtype or high eIF4E expression.
* ECOG performance status 0, 1, 2 or 3.
* Life expectancy > 4 weeks.
* Age is > 18 years.
* Female patients of childbearing potential must have a negative serum (beta-HCG) pregnancy test within 14 days of starting protocol and must not be breastfeeding. Men and women of childbearing potential must agree to use an effective means of contraception throughout the study and for at least 30 days after completion of protocol.
* Adequate renal and hepatic function: serum creatinine < 1.5 x ULN; AST or ALT < 2.5 x ULN (or < 5 x ULN if liver involvement with leukemia); serum bilirubin < 1.5 x ULN.
* Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.
* Accessible for treatment and follow up.

Exclusion Criteria:

* Uncontrolled central nervous system involvement by AML.
* Active cardiovascular disease as defined by New York Heart Association (NYHA) class III-IV categorization.
* Intercurrent illness or medical condition precluding safe administration of the planned protocol treatment or required follow-up.
* Received any previous therapy for AML within 28 days prior to the study entry. Hydrea is permitted for the treatment of leukocytosis but must be stopped within 7 days of starting low dose ara-C and ribavirin.
* Female patients who are pregnant or breastfeeding.
* Concurrent treatment with other anti-cancer therapy.
* Known infection with HIV.
* History of other malignancy. Subjects who have been disease-free for 2 year or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* FAB AML M1, 2, 6, 7 will be excluded if they do not have high eIF4E expression. AML M3 is always excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Assouline, MD, Principal Investigator — Jewish General Hospital, McGill University; Katherine Borden, PhD, Study Director — Université de Montréal
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Assouline S, Culjkovic B, Cocolakis E, Rousseau C, Beslu N, Amri A, Caplan S, Leber B, Roy DC, Miller WH Jr, Borden KL. Molecular targeting of the oncogene eIF4E in acute myeloid leukemia (AML): a proof-of-principle clinical trial with ribavirin. Blood. 2009 Jul 9;114(2):257-60. doi: 10.1182/blood-2009-02-205153. Epub 2009 May 11. PMID 19433856
- [Result] Assouline S, Culjkovic-Kraljacic B, Bergeron J, Caplan S, Cocolakis E, Lambert C, Lau CJ, Zahreddine HA, Miller WH Jr, Borden KL. A phase I trial of ribavirin and low-dose cytarabine for the treatment of relapsed and refractory acute myeloid leukemia with elevated eIF4E. Haematologica. 2015 Jan;100(1):e7-9. doi: 10.3324/haematol.2014.111245. Epub 2014 Nov 25. No abstract available. PMID 25425688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in this dose escalation study according to a 3+3 design. Patients not completing 28 days of therapy were replaced as they were not evaluable for the pharmacokinetic endpoint of steady state level of ribavirin.
Groups:
- Dose Level 1: Ribavirin 1000 mg po bid x 28 days, cytarabine arabinoside 20 mg sc bid days 1 to 10
- Dose Level 2: Ribavirin 1400 mg po bid x 28 days, cytarabine arabinoside 20 mg sc bid days 1 to 10
- Dose Level 3: Ribavirin 1800 mg po bid x 28 days, cytarabine arabinoside 20 mg sc bid days 1 to 10
- Dose Level 4: Ribavirin 2200 mg po bid x 28 days, cytarabine arabinoside 20 mg sc bid days 1 to 10
- Dose Level 5: Ribavirin 1000 mg po bid x 28 days, cytarabine arabinoside 10 mg sc bid days 1 to 10
- Dose Level 6: Ribavirin 1400 mg po bid x 28 days, cytarabine arabinoside 10 mg sc bid days 1 to 10
- Dose Level 7: Ribavirin 1800 mg po bid x 28 days, cytarabine arabinoside 10 mg sc bid days 1 to 10
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Dose Level 7
Started | 4 | 3 | 5 | 6 | 3 | 3 | 5
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 4
Not Completed | 1 | 0 | 2 | 3 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 2 | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ribavirin and Cytarabine: Dose level 1 = 1000 mg po BID/ Dose level 2 = 1400 mg po BID/ Dose level 3 = 1800 mg po BID Drug: Cytarabine arabinoside Previous cohorts at 20 mg bid days 1 to 10 of every 28 day cycle. Dosage modified to 10 mg bid days 1 to 10 of every 28 day cycle for more recent cohorts.
Arm/Group | Ribavirin and Cytarabine
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 65 [22 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
FAB subtype [Count of Participants; unit: Participants] — FAB - French American British leukemia classification
  Participants
    FAB sutype M4/M5 | 22
    Other FAB subtypes | 7

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RP2D) of Ribavirin When Given in Combination With Low-dose Ara-C
Description: This 3+3 designed aimed to determine recommended phase II dose (RP2D) based on pharmacokinetics (PK) and maximum tolerated dose (MTD). For the dose to be selected, a target steady state level of ribavirin 20 uM was needed for all patients and no more than 1 of 6 patients could have had dose limiting toxicity at that dose.
Time Frame: 56 days
Measure: Number; unit: mg
Groups:
- Ribavirin-Cytarabine: Ribavirin: Dose level 1 = 1000 mg po BID/ Dose level 2 = 1400 mg po BID/ Dose level 3 = 1800 mg po BID
  Cytarabine arabinoside: Previous cohorts at 20 mg bid days 1 to 10 of every 28 day cycle.
  Dosage modified to 10 mg bid days 1 to 10 of every 28 day cycle for more recent cohorts.
Arm/Group | Ribavirin-Cytarabine
Number analyzed (Participants) | 29
mg
  Ribavirin po bid for 28 days | 1400
  cytarabine arabinoside sc bid for 10 days | 10

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate comprises complete response (<5% blasts in the bone marrow, and in the peripheral blood Hgb more than or equal to 100 g/L, platelets more than or equal to 100x10-9/L, and neutrophils more than or equal to 1x10-9/L), partial response (5 to 25% blasts in the bone marrow and same peripheral blood parameters) and blast response (a greater than 50% decrease in bone marrow blast count and 2 log reduction in peripheral blood blast count, sustained for at least 28 days).
Time Frame: 2-3 years
Population: Only patients treated for 28 days or more were evaluable for response.
Measure: Count of Participants; unit: Participants
Groups:
- Ribavirin and Cytarabine: Patients with relapsed or refractory AML or elderly untreated AML with FAB subtype M4/M5 or overexpressing eIF4E were treated with ribavirin and cytarabine arabinoside according to a 3+3 dose escalation scheme
Arm/Group | Ribavirin and Cytarabine
Number analyzed (Participants) | 21
Participants | 5

3. Secondary Outcome: Complete Response Rate
Description: Defined as <5% blasts in the bone marrow and a hgb 100 g/L, platelets 100,000/uL, neutrophils 1000/uL.
Time Frame: 2-3 years
Population: Only patients treated for at least 28 days were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribavirin and Cytarabine
Number analyzed (Participants) | 21
Participants | 2

4. Secondary Outcome: Partial Response
Description: Partial response was defined as 5 to 25% blasts in the bone marrow and Hgb >100g/L, platelets >100,000/ul and neutrophils >1000/ul.
Time Frame: 2-3 years
Population: Only patients treated for 28 days or more were assessed for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribavirin and Cytarabine
Number analyzed (Participants) | 21
Participants | 1

5. Secondary Outcome: Blast Response
Description: Blast response was defined as a greater than 50% decrease in bone marrow blast count and 2 log reduction in peripheral blood blast count, sustained for at least 28 days.
Time Frame: 2-3 years
Population: Only patients treated for 28 days or more were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribavirin and Cytarabine
Number analyzed (Participants) | 21
Participants | 2

ADVERSE EVENTS:
Time Frame: 44 months
Arm/Group | Ribavirin-Cytarabine
Serious Adverse Events (participants affected / at risk) | 7/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin-Cytarabine (N=29)
Syncope (Nervous system disorders) | 1
Exacerbation of bone pain (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular hemorrhage (Nervous system disorders) | 1
retinal hemorrhage (Eye disorders) | 1
visceral shingles (Infections and infestations) | 1
Lower gastro-intestinal hemorrhage (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin-Cytarabine (N=29)
Hemolytic Anemia (Blood and lymphatic system disorders) | 4
anorexia (Gastrointestinal disorders) | 3
nausea (Gastrointestinal disorders) | 7
diarrhea (Gastrointestinal disorders) | 5
mucositis (Gastrointestinal disorders) | 12
vomiting (Gastrointestinal disorders) | 6
dry mouth (Gastrointestinal disorders) | 2
low potassium (Metabolism and nutrition disorders) | 4
high ALT (Investigations) | 4
anemia (Blood and lymphatic system disorders) | 15
neutropenia (Blood and lymphatic system disorders) | 5
thrombocytopenia (Blood and lymphatic system disorders) | 7
fatigue (General disorders) | 12
fever (General disorders) | 6
high bilirubin (Investigations) | 2
chills (General disorders) | 2
high uric acid (Investigations) | 2
dizziness (Nervous system disorders) | 2
infection (Infections and infestations) | 8
febrile neutropenia (Blood and lymphatic system disorders) | 13
pneumonia (Infections and infestations) | 3
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
headache (Nervous system disorders) | 2
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2
generalized weakness (Musculoskeletal and connective tissue disorders) | 5
muscle cramps (Musculoskeletal and connective tissue disorders) | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
cough (Respiratory, thoracic and mediastinal disorders) | 3
rash (Skin and subcutaneous tissue disorders) | 2
hematoma (Vascular disorders) | 2
petechia (Blood and lymphatic system disorders) | 5

LIMITATIONS AND CAVEATS:
There were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No